CLINICAL TRIAL: NCT03291717
Title: Randomized Trial of a Peer-led Intervention to Promote Community Living and Participation - The Bridging Community Gaps Photovoice
Brief Title: Bridging Community Gaps Photovoice
Acronym: BCGP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Mental Health Center of Denver (Unknown); Connecticut State, Department of Mental Health and Addiction Services (Other Government); Riverside Community Care (Unknown)
Responsible Party: Principal Investigator, Erna Sally Rogers, Research Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4591
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Mental Illness; Social Isolation
Keywords: Mental Illness; Community Participation; Stigma; Photovoice
MeSH Terms: conditions — Mental Disorders; Social Isolation; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bridging Community Gaps Photovoice (BCGP) (Experimental): The BCGP program is a 6-month photovoice-based intervention to help individuals with psychiatric disabilities enhance their community participation.
  Interventions: Behavioral: Bridging Community Gaps Photovoice (BCGP)
- Services as Usual (No Intervention): Individuals in this group continue with their regular mental health services with no additional intervention.

INTERVENTIONS:
Behavioral: Bridging Community Gaps Photovoice (BCGP) — Participants assigned to this group will be part of the 6-month long BCGP intervention, which involves a 12- week class that meets weekly, followed by three booster sessions - one per month in the three months following the class, and up to 24 sessions of individual support as needed throughout the 6 months provided on a weekly basis either in person or by phone. The BCGP classes follow a manualized curriculum with sessions that combine didactic information, Photovoice exercises, and group discussions to empower participants in pursuing community participation goals, all refined with input from individuals with a lived experience.
  Arms: Bridging Community Gaps Photovoice (BCGP)

SUMMARY:
The purpose of this study is to test a peer-led intervention intended to promote the community living and participation of individuals with psychiatric disabilities entitled "Bridging Community Gaps Photovoice" (BCGP). The intervention targets increasing community involvement of individuals with psychiatric disabilities through reduction in self-stigma and perceived stigma, enhancing opportunities for community participation, and support to achieve community participation goals.

DETAILED DESCRIPTION:
The BCGP intervention is 6 months long and the investigators expect that participants will experience lower self and perceived stigma, increased community participation and sense of belonging, and improved psychosocial functioning and personal growth after the intervention. The intervention is comprised of a 12-week class that meets once a week for two hours, followed by three booster sessions - one per month in the three months following the class, and up to 24 sessions of individual support as needed throughout the 6 months provided on a weekly basis either in person or by phone. The purpose of the individual support is to reinforce the class activities and to ensure the participants meets their community participation goal. The proposed study is a randomized trial which will be conducted at Boston University Center for Psychiatric Rehabilitation (BUCPR) in Massachusetts, the Mental Health Center of Denver (MHCD) in Colorado, and the Greater Bridgeport Mental Health Center (GBMHC) in Connecticut.

ELIGIBILITY:
Inclusion Criteria:

1. are 18 or older.
2. are recipients of services at research sites due to having a DSM-V diagnosis of mental illness, including dual diagnosis (dual diagnosis refers to co-occurring mental illness and alcohol/ substance use disorder).
3. are interested in enhancing their community participation.
4. are not currently receiving individual peer support services.
5. are able to read and write in English.

Exclusion Criteria:

1)Inability to give full and knowing consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
UCLA Loneliness Scale | Change from Baseline to 3 months to 6 months to 9 months to 12 months
  is a 20-item 4-point Likert-type scale, widely used measure of loneliness and social isolation. Cronbach's alpha coefficients ranging from .89 to .94.
Multi-Dimensional Assessment of Community Participation | Change from Baseline to 3 months to 6 months to 9 months to 12 months
  Consists of a set of objective and subjective measures of community belonging, inclusion and participation.

SECONDARY OUTCOMES:
Internalized Stigma of Mental Illness Scale | Change from Baseline to 3 months to 6 months to 9 months to 12 months
  29-item, 4-point scale from (strongly disagree to strongly agree) assesses behaviors, thoughts and feelings that are self-stigmatizing including alienation, stereotype endorsement, social withdrawal, stigma resistance.
The Stigma Scale | Change from Baseline to 3 months, 3 months to 6 months, 6 months to 9 months, 9 months to 12 months
  28 item, 5 point scale (strongly disagree to strongly agree) measuring experienced and anticipated stigma.
Approaches to Coping with Anti-Stigma | Change from Baseline to 3 months to 6 months to 9 months to 12 months
  27-item instrument with a 4 point scale (strongly disagree to strongly agree) measuring strategies to cope with stigma: secrecy, withdrawal, educating, challenging, and distancing.
Personal Growth and Recovery Scale | Change from Baseline to 3 months to 6 months to 9 months to 12 months
  25-item, 4 point scale (strongly disagree to strongly agree) of items measuring psychosocial functioning and recovery.
Community Goal Achievement Scale | Change from Baseline to 3 months to 6 months to 9 months to 12 months
  adapted from Goal Attainment Scale, provides a structured approach to determining goal achievement regardless of the type or uniqueness of goal .
Behavior and Symptom Identification Scale (BASIS - R) | Change from Baseline to 3 months to 6 months to 9 months to 12 months
  A 24-item scale that measures: mood disturbances, anxiety, interpersonal and role functioning, daily living skills, psychotic symptoms, impulsivity and substance use

CONTACTS AND LOCATIONS:
Overall Officials: Erna S Rogers, PhD, Principal Investigator — Boston University
Locations (4):
- United States (4):
  - Mental Health Center of Denver, Denver, Colorado
  - Greater Bridgeport Mental Health Center, Bridgeport, Connecticut
  - Boston University, Center for Psychiatric Rehabilitation, Boston, Massachusetts
  - Horizon House- Riverside Community Care, Wakefield, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided